CLINICAL TRIAL: NCT05971069
Title: Real-time Identification of the Aberrant Left Hepatic Arterial Territory in the Liver Using Near-infrared Fluorescence Imaging: Prospective Study to Develop Decision Algorithm to Define the Preservation/Ligation of an Aberrant Left Hepatic Artery
Brief Title: Real-time Identification of the Aberrant Left Hepatic Arterial Territory in the Liver Using Near-infrared Fluorescence Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Associate Professor, Gangnam Severance Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2021-0376
Record Dates: First submitted 2023-07-04; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Masking Description: Enrolled patients will be divided into three groups according to the real time near-infrared fluorescence imaging during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1 (Experimental): Entire fluorescence defect on the Lt. lobe of liver → Preservation of the aberrant left hepatic artery
  Interventions: Procedure: Group1
- Group2 (Experimental): Partial fluorecence defect on the Lt. lobe of liver → Ligation of the aberrant left hepatic artery
  Interventions: Procedure: Group2
- Group3 (Experimental): No fluorescence defect on the Lt. lobe of liver → Ligation of the aberrant left hepatic artery
  Interventions: Procedure: Group3

INTERVENTIONS:
Procedure: Group1 — Entire fluorescence defect on the Lt. lobe of liver → Preservation of the aberrant left hepatic artery
  Arms: Group1
Procedure: Group2 — Partial fluorecence defect on the Lt. lobe of liver → Ligation of the aberrant left hepatic artery
  Arms: Group2
Procedure: Group3 — No fluorescence defect on the Lt. lobe of liver → Ligation of the aberrant left hepatic artery
  Arms: Group3

SUMMARY:
" Hepatic artery variants are occasionally seen, especially 20-30% of aberrant left hepatic artery. In radical gastrectomy, decision for aberrant left hepatic artery(ALHA) ligation should consider the oncologic safety and liver-related complication. Theoretically, the ALHA preservation is the most ideal in the aspect of liver function protection. However, it is technically difficult which consumes much time. Not only that, oncologic safety could be threatened as some soft tissues, including lymph nodes, could be remained while in preserving the ALHA.

There has been no standardized method to evaluate the ALHA, and to decide whether preserve or ligate it.

This prospective study has been designed to develop the decision algorithm to define the ALHA preservation/ligation, using near-infrared fluorescence imaging during surgery. "

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with gastric adenocarcinoma pathologically before surgery
2. Patients aged between 20 to 80
3. Patients with an ECOG 0 or 1
4. Patients who were confirmed the presence of aberrant left hepatic artery before or during surgery

Exclusion Criteria:

1. Patients with abnormal liver function test befor surgery
2. Patients who diagnosed liver cirrhosis or infectious liver disease
3. Patients who underwent liver resection, or chemotherapy for gastric cancer
4. Patients planned for combined liver resection or cholecystectomy during gastrectomy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
The safety and efficacy of the decision algorithm for the aberrant left hepatic artery preservation/ligation with real time near-infrared fluorescence imaging | Real time near-infrared fluorescence image will be obtained during the surgery.
  Investigator discretionally designed the decision algorithm for aberrant left hepatic artery preservation/ligation with real time near-infrared fluorescence imaging.
  The order of the algorithm is as follows:
  First, when surgeons identify the aberrant left hepatic artery during surgery, clamping the artery and injectioning indocyanine green (5mg/mL) intravenously would be performed.
  After that, in a few seconds, liver perfusion could be detected through real time near-infrared fluorescence imaging.
  The ligation or preservation of the aberrant left hepatic artery would be decided according to the proportion of the near-infrared fluorescence imaging defect. Investigator's like to confirm the safety and efficacity of this decision algorithm.

SECONDARY OUTCOMES:
Number of participants with liver-related postoperative complications as assessed by serum aspartate transaminase(AST) and alanine transferase(ALT) | Serum aspartate transaminase(AST, IU/L) and alanine transferase(ALT, IU/L) will be estimated in postoperative 1st, 2nd, 3rd and 5th day.
  The elevated proprtion of the serum aspartate transaminase(AST, IU/L) and alanine transferase(ALT, IU/L) compared to preoperative value will be calculated and compared by groups.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea